CLINICAL TRIAL: NCT03479814
Title: AIDA-RE-1: Adaptive Individualized Hig-Dose Radiotherapy Analysis-Rectum-1. Interventional Study on Neoadjuvant Adaptive-treatment of High Risk Rectal Cancer
Brief Title: Adaptive Individualized High-Dose Radiotherapy Analysis-REctum-1 (AIDA-RE-1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIDA-RE-1
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Rectal Cancer; Radiotherapy; Neoadjuvant Treatment
Keywords: rectal cancer; neoadjuvant chemoradiation; IMRT-SIB; adaptive radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMRT-SIB plus sequential IG-RT boost (Experimental): 45 Gy plus 5 Gy concomitant boost are delivered to rectum and locoregional lymphnodes (25 fractions); sequential IG-RT (imaging guided-radiotherapy) boost of 5 Gy in 2 fractions is planned with 18-FDG-PET
  Interventions: Radiation: IMRT-SIB plus sequential IG-RT boost

INTERVENTIONS:
Radiation: IMRT-SIB plus sequential IG-RT boost

SUMMARY:
Aim of the study is to evaluate achievement of complete pathologic response (pCR) in high-risk rectal cancer treated with neoadjuvant concomitant chemotherapy plus adaptive-intensity modulated imaging-guided radiotherapy

DETAILED DESCRIPTION:
AIDA-RE-1 is an interventional prospective trial for the treatment of locally advanced high-risk rectal cancer. In neoadjuvant setting, patients are treated with standard chemotherapy plus experimental radiotherapy. The total dose to clinical target volume (CTV, rectum and locoregional lymph nodes) is 45 Gy, with a concomitant boost of 5 Gy to gross tumor volume (GTV), delivered with IMRT-SIB (intensity modulated radiotherapy-simultaneous integrated boost) technique in 25 fractions. After 2 weeks of treatment, patients are evaluated with 18 FDG-PET and sequential boost of 5 Gy (in 2 fractions) is planned.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of locally advanced rectal cancer (cT3N+, cT4Nx, local relapse, cT3N0); cT2N+ is acceptable if low rectum is involved
* M0
* ECOG 0-2

Exclusion Criteria:

* M1
* familial adenomatous polyposis (FAP), non-polyposis hereditary colorectal cancer, inflammatory bowel disease
* severe cardiopathy
* previous pelvic RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2016-08-01; Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
complete pathological response (pCR) | 6 weeks
  pCR is defined as ypT0N0

SECONDARY OUTCOMES:
Acute toxicity | 6 months
  Acute toxicity is evaluated using CTCAE criteria
Quality of Life (QoL) | 1 year
  QoL is evaluated using EORTC QoL questionnaire
Late toxicity | 1 year
  Late toxicity is evaluated using CTCAE criteria
Dosimetric advantage of GTV-boost reduction | 6 weeks
  Dosimetric advantage is evaluated using DVHs (Dose Volume Histograms)
Evaluation of PET-response as predictive factor | 1 year
  Correlation between SUV (Standardized Uptake Value) and pathological response

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, Unversity of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy
Locations (1):
- Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine- DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No